CLINICAL TRIAL: NCT05868512
Title: Effectiveness of Dry Needling Versus Therapeutic Ultrasound Along With Routine Physical Therapy in Patients With for Chronic Neck Pain; a Randomized Control Trial
Brief Title: Effectiveness of DN Versus TU Along With Routine PT in Patients With for Chronic Neck Pain RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/528
Record Dates: First submitted 2023-03-18; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Other)
  Interventions: Diagnostic Test: Dry needling
- therapeutic ultrasound (Experimental)
  Interventions: Diagnostic Test: Therapeutic ultrasound

INTERVENTIONS:
Diagnostic Test: Dry needling — Dry Needling Along With Routine Physical Therapy for Chronic Neck Pain
  Arms: Dry needling
Diagnostic Test: Therapeutic ultrasound — Therapeutic ultrasound Along With Routine Physical Therapy for Chronic Neck Pain
  Arms: therapeutic ultrasound

SUMMARY:
To determine the effectiveness of dry needling and therapeutic ultrasound for the treatment of chronic neck pain

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be office workers having pain sensation at neck for at least 4 months
* pain for 3-7 on NRS and with the limited or painful ROM.
* Age of the participants will be 20-35 years.
* Only those individuals will be included who are working in the field for more than 8 months and work for 6-8 hours per day.

Exclusion Criteria:

* The exclusion criteria were any other neurological conditions of cervical vertebra, cervical radiculopathy, any vascular disease, tumors or any other local infection

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Range of Motion Scale | 3 Months
  Range of Motion is a measuring scale, specifically designed to allow patients and providers to measure the opening, movement and function of the mouth and jaw
Visual Analog Scale for pain the lower score is better | 3 Months
  Visual Analog Scale Ranges1-10 scaling normal to worst

CONTACTS AND LOCATIONS:
Locations (1):
- Households, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No